CLINICAL TRIAL: NCT01327742
Title: Phase II Clinical Study of the Safety and Efficacy of the Relay Thoracic Stent-Graft in Patients With Thoracic Aortic Pathologies
Brief Title: Phase II Clinical Study of the Safety and Efficacy of the Relay Thoracic Stent-Graft
Status: Approved for marketing | Type: Expanded Access
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IP-0004-06 rev I
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Thoracic Aortic Aneurysm; Penetrating Ulcers
Keywords: Relay; Thoracic; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer; Aneurysm

INTERVENTIONS:
Device: Relay Thoracic Stent-Graft — Device implant

SUMMARY:
This study is a continuation of the pivotal trial studying the safety and efficacy of the Relay thoracic stent-graft system to treat thoracic aortic aneurysms. Efficacy is being evaluated by the device-related adverse event rate of endovascular repair (via the Relay thoracic stent-graft) through 1 year. Safety is being evaluated by comparing major adverse events through 1 year in subjects treated with the Relay thoracic stent-graft to those who underwent surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed descending thoracic aneurysm or penetrating ulcer
* Subjects whose anatomy can accommodate the Relay device
* Subjects who consent to participate
* Subjects who agree to a follow-up schedule

Exclusion Criteria:

* Subjects with lesions other than thoracic aneurysm and penetrating ulcer
* Subjects with less than 1 year life expectancy
* Subjects who are pregnant
* Subjects with medical conditions that wold complicate the endovascular procedure or confound results (e.g., Marfan's syndrome, morbid obesity, severe coronary artery disease)
* Subjects participating in another investigational study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Arizona Heart Hospital, Phoenix, Arizona
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Sentara Heart Hospital, Norfolk, Virginia
  - University Washington, Seattle, Washington